CLINICAL TRIAL: NCT01417273
Title: Impact of Vitamin A Supplementation on Disease Activity and Progression in Multiple Sclerotic (MS) Patients
Brief Title: Impact of Vitamin A on Multiple Sclerosis (MS)
Acronym: MS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Ali Akbar Saboor-Yaraghi/ Assistant professor, Tehran University of Medical Sciences(TUMS)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8887
Record Dates: First submitted 2010-11-17; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; immune system; vitamin A; (MSFC)Multiple Sclerosis Functional Composite; (EDSS)Expanded Disability Status Scale; (MRI)Magnetic resonance imaging
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin A, multiple sclerosis, (Active Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 25000 IU/day vitamin A for 6 months and 10000 IU/day for next 6 months
  Interventions: Dietary Supplement: vitamin A; Drug: Drug: placebo
- placebo/Multiple Sclerosis (Placebo Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 1 cap of placebo/day
  Interventions: Dietary Supplement: vitamin A

INTERVENTIONS:
Dietary Supplement: vitamin A — 1 cap vitamin A 25000 IU/day for 6 months and 10000 IU/day for next 6 months
Drug: Drug: placebo — 1 cap placebo/day for 12 month
  Arms: vitamin A, multiple sclerosis,

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with 25000 IU preformed vitamin A (retinyl palmitate) or placebo for first 6 months and 10000 IU/day for next 6 months on disease activity and progression in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease where Th1 like responses from myelin-specific CD4+ T cells, as secretion of pro-inflammatory IFNγ, are believed to play a major role in the pathogenesis. The myelin-specific T cells that mediate tissue destruction in MS are believed to become activated outside the central nervous system (CNS) in lymphoid tissue and when they cross the blood brain barrier they will re-encounter their antigen. Immune deviation is the redirection of the immune response from most often Th1 like responses to Th2 like responses, even though the opposite can also occur. Vitamin A or Vitamin A-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. High level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid(RA) inhibits IL12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or RA decreases IFNγ and increases IL5, IL10, and IL4 production.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have used interferon beta in last 3 months
* Patients with 0-5 EDSS

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR

  * Patients who have allergy to vitamin A compounds, OR
  * Patients who have used vitamin supplements in last 3 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Change from baseline at 12 months
  Expanded Disability Status Scale (EDSS) as a measure of activity and progression of MS disease
Multiple Sclerosis Functional Composite (MSFC) | Change from baseline at 12 months
  Multiple Sclerosis Functional Composite (MSFC) as a measure of activity and progression of MS disease
fatigue scores | Change from baseline at 12 months
  fatigue scores on Multiple Sclerosis Fatigue Impact Scale
depression score | Change from baseline at 12 months
  depression score on Beck Depression Inventory 2
Number of active lesion in magnetic resonance imaging (MRI) number of active lesion in brain MRI | Change from baseline at 12 months
  Number of active lesion in magnetic resonance imaging (MRI) as a measure of activity and progression of MS disease

SECONDARY OUTCOMES:
number of disease relapses | Change from baseline at 12 months
  To measure the effect of vitamin A supplementation on number of disease relapses

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akbar saboor Yaraghi, PhD, Study Chair — Tehran University of Medical Sciences; Sama Bitarafan, MD, PhD student, Principal Investigator — Tehran University of Medical Siences
Locations (1):
- Tehran University of Medical Sciences,, Tehran, Iran

REFERENCES:
- [Derived] Bitarafan S, Saboor-Yaraghi A, Sahraian MA, Soltani D, Nafissi S, Togha M, Beladi Moghadam N, Roostaei T, Mohammadzadeh Honarvar N, Harirchian MH. Effect of Vitamin A Supplementation on fatigue and depression in Multiple Sclerosis patients: A Double-Blind Placebo-Controlled Clinical Trial. Iran J Allergy Asthma Immunol. 2016 Feb;15(1):13-9. PMID 26996107
- [Derived] Bitarafan S, Saboor-Yaraghi A, Sahraian MA, Nafissi S, Togha M, Beladi Moghadam N, Roostaei T, Siassi F, Eshraghian MR, Ghanaati H, Jafarirad S, Rafiei B, Harirchian MH. Impact of Vitamin A Supplementation on Disease Progression in Patients with Multiple Sclerosis. Arch Iran Med. 2015 Jul;18(7):435-40. PMID 26161708